CLINICAL TRIAL: NCT02978430
Title: Implementation of Computer-Assisted Intraoperative Goal-Directed Fluid Therapy in Major Abdominal Surgery: A Before and After Study
Brief Title: Implementation of Computer-Assisted Intraoperative Goal-Directed Fluid Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Prevention
Other Study IDs: P2016/334
Record Dates: First submitted 2016-11-22; First posted 2016-12-01 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2016-11

CONDITIONS: Major Abdominal Surgery
Keywords: Fluid therapy; Anesthesiology; Major surgery; Goal-directed fluid therapy; Fluid responsiveness; Closed-loop system
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (Active Comparator): This group (started retrospectively before the first included patient of the closed-loop goal-directed fluid therapy group) consists of patients undergoing major abdominal surgery where fluid management is carried out based only on static variables (e.g. arterial pressure, heart rate, CVP, and urine output).
  Interventions: Other: Standard of care
- Computer-assisted GDFT (Active Comparator): This group consists of patients undergoing major abdominal surgery where fluid management is carried out with a closed-loop (automated) system to deliver fluid by a goal-directed fluid therapy (GDFT) standardized protocol.
  Confer: "Crystalloids or Colloids for Goal-directed Fluid Therapy With Closed-loop Assistance in Major Surgery" (NCT02312999)
  Interventions: Device: Computer-assisted GDFT

INTERVENTIONS:
Device: Computer-assisted GDFT — Patients receive fluid therapy via a computer-assisted goal-directed fluid therapy (GDFT) prototype closed-loop (automated) system guided by a cardiac output monitor.
  Arms: Computer-assisted GDFT
Other: Standard of care — Patients receive fluid management based only on static variables (e.g. arterial pressure, heart rate, CVP, and urine output). This control group (started retrospectively before the first included patient of the closed-loop goal directed fluid therapy group) consists of the same population undergoing the same surgery as the closed-loop GDFT group.
  Arms: Standard of care

SUMMARY:
The aim of this study is to compare the implementation of computer-assisted goal directed fluid therapy (GDFT) to standard of care fluid therapy in major abdominal surgery.

DETAILED DESCRIPTION:
Fluid therapy is one of the main tools used in anesthesiology to maintain adequate hemodynamic stability. Goal-directed fluid therapy (GDFT) based on cardiac output and/or dynamic parameters of fluid responsiveness (e.g. pulse pressure variation) has been shown to decrease post-operative complications. The main inconvenience of protocol based therapy is its technical complexity which requires considerable time, attention, and vigilance. GDFT assisted by a closed-loop system, when compared to manual GDFT, is associated with a longer preload independent state and could increase clinician adherence to protocol. To this day no study has compared closed-loop assisted GDFT to standard of care.

Goal:

This study compares the results of the study entitled "Crystalloids or Colloids for Goal directed Fluid Therapy With Closed-loop Assistance in Major Surgery" (NCT02312999) to a standard of care group (started retrospectively before the first included patient of the above study) where fluid therapy is based only on static variables (e.g. arterial pressure, heart rate, central venous pressure (CVP), and urine output.) These groups consisted of the same population undergoing the same types of surgery.

Hypothesis:

A protocolized approach using computer-assisted GDFT when compared to standard of care is associated with less fluid administration and less blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over the age of 18) undergoing elective major abdominal surgery that is expected to take longer than 3 hours and requiring general anesthesia.

Exclusion Criteria:

* Patients under 18 years of age
* Patients not undergoing surgery, requiring anesthesia, or cardiac output monitoring
* Patients with arrhythmia and/or atrial fibrillation
* Patients who are allergic to HES (hydroxyethyl starch)
* Patients with renal insufficiency (serum creatinine of >2 mg/ml) or hepatic dysfunction (liver enzymes >1.5)
* Patients who has coagulation disorders (values higher than 1.5x normal values)
* Patients without the capacity to give written informed consent or refusal of consent
* Pregnancy at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Perioperative fluid administration | 24 hours
  Fluid balance during perioperative period

SECONDARY OUTCOMES:
Length of hospitalisation | Every day up to 90 days after hospitalization
Mortality rate | 30 days
Transfusion of blood products during hospitalization | Every day up to 90 days post surgery
  In-hospital transfusion during hospitalization
Hypotension incidence during surgery | 24 hours
  Incidence of hypotension (defined as total case time spent with 20% drop from baseline preoperative blood pressure)
Need of vasopressor | 24 hours
  Use of vasopressors during the perioperative period
Renal function - urea level | Every day up to 90 days after hospitalization
  Urea levels. Measured in a blood sample taken during hospitalization
Renal function - creatinine level | Every day up to 90 days after hospitalization
  Creatinine levels. Measured in a blood sample taken during hospitalization
Postoperative complications | Every day up to 90 days after hospitalization
  Major complications included cardiac (acute coronary syndrome/ arrhythmia), pulmonary (embolism/edema), gastrointestinal (bowel and surgical anastomotic leak/internal or external fistulas/peritoneal effusions), renal (renal failure requiring dialysis), infectious (peritonitis/ sepsis), coagulation (bleeding), wound dehiscence, stroke, reoperation, readmission, and death. Minor complications included unplanned ICU admission, pneumonia/pleural effusion, deep venous thrombosis, paralytic ileus progressive, renal insufficiency, infection (superficial wound infection/fever/urinary infection) and confusion/delirium.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scheeren TW, Wiesenack C, Gerlach H, Marx G. Goal-directed intraoperative fluid therapy guided by stroke volume and its variation in high-risk surgical patients: a prospective randomized multicentre study. J Clin Monit Comput. 2013 Jun;27(3):225-33. doi: 10.1007/s10877-013-9461-6. Epub 2013 Apr 5. PMID 23558909
- [Background] Salzwedel C, Puig J, Carstens A, Bein B, Molnar Z, Kiss K, Hussain A, Belda J, Kirov MY, Sakka SG, Reuter DA. Perioperative goal-directed hemodynamic therapy based on radial arterial pulse pressure variation and continuous cardiac index trending reduces postoperative complications after major abdominal surgery: a multi-center, prospective, randomized study. Crit Care. 2013 Sep 8;17(5):R191. doi: 10.1186/cc12885. PMID 24010849
- [Background] Spanjersberg WR, Bergs EA, Mushkudiani N, Klimek M, Schipper IB. Protocol compliance and time management in blunt trauma resuscitation. Emerg Med J. 2009 Jan;26(1):23-7. doi: 10.1136/emj.2008.058073. PMID 19104091
- [Background] Rinehart J, Lilot M, Lee C, Joosten A, Huynh T, Canales C, Imagawa D, Demirjian A, Cannesson M. Closed-loop assisted versus manual goal-directed fluid therapy during high-risk abdominal surgery: a case-control study with propensity matching. Crit Care. 2015 Mar 19;19(1):94. doi: 10.1186/s13054-015-0827-7. PMID 25888403
- [Derived] Joosten A, Coeckelenbergh S, Delaporte A, Ickx B, Closset J, Roumeguere T, Barvais L, Van Obbergh L, Cannesson M, Rinehart J, Van der Linden P. Implementation of closed-loop-assisted intra-operative goal-directed fluid therapy during major abdominal surgery: A case-control study with propensity matching. Eur J Anaesthesiol. 2018 Sep;35(9):650-658. doi: 10.1097/EJA.0000000000000827. PMID 29750699